CLINICAL TRIAL: NCT03882762
Title: A Non-randomized, Single-dose, Open-Label, Pharmacokinetic Study of Cebranopadol in Patients With Impaired Renal Function and Subjects With Normal Renal Function
Brief Title: A Clinical Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of Cebranopadol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GRT-PK-07
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Pharmacokinetic
MeSH Terms: interventions — 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group I - Cebranopadol 200 μg tablet (Experimental): Mild Renal Impairment:
  PK evaluable non-dialyzed patients with mildly impaired renal function (eGFR = 60-89 mL/min/1.73 m2)
  Interventions: Drug: Cebranopadol 200 μg tablet
- Group II - Cebranopadol 200 μg tablet (Experimental): Moderate Renal Impairment:
  PK evaluable non-dialyzed patients with moderately impaired renal function (eGFR = 30-59 mL/min/1.73 m2)
  Interventions: Drug: Cebranopadol 200 μg tablet
- Group III - Cebranopadol 200 μg tablet (Experimental): Severe Renal Impairment:
  PK evaluable non-dialyzed patients with severely impaired renal function (eGFR = 15-29 mL/min/1.73 m2)
  Interventions: Drug: Cebranopadol 200 μg tablet
- Group IV - Cebranopadol 200 μg tablet (Experimental): Normal Renal Function:
  PK evaluable participants with normal renal function (eGFR greater than or equal to 90 mL/min/1.73 m2)
  Interventions: Drug: Cebranopadol 200 μg tablet

INTERVENTIONS:
Drug: Cebranopadol 200 μg tablet — 200 μg cebranopadol film-coated tablet was taken with 240 mL of water under fed conditions.

SUMMARY:
The objective of this study was to evaluate the pharmacokinetics (PK), safety and tolerability profile of cebranopadol (GRT6005) in patients with varying degree of renal impairment and participants with normal renal function after an oral single dose administration.

This study was a Phase 1, multi-center, non-randomized, open-label, parallel group, single-dose study in up to 24 male and female patients with varying degree of renal impairment and participants with normal renal function.

Within 14 days before the administration of cebranopadol the general eligibility of the participants for the study was assessed according to the inclusion/exclusion criteria. Estimated glomerular filtration rate (eGFR) was determined according to the Modification of Diet in Renal Disease (MDRD) equation.

A treatment period from Day -1 to Day 8 was performed, with participant confinement to the study site from Day -1 to Day 6 and an outpatient visit on Day 8. A single dose of cebranopadol 200 μg was administered on Day 1. Multiple blood and urine samples were drawn for pharmacokinetic evaluations and safety laboratory monitoring. Additional blood samples were taken prior investigational medicinal product (IMP) administration to assess serum creatinine concentration and protein binding.

An End-of-Trial Visit was performed at the time, or within 7 days, of the final blood sample on Day 8 or at early withdrawal.

ELIGIBILITY:
Inclusion Criteria:

Common criteria:

* Sign the informed consent form (ICF) and have the mental capability to understand it.
* Be male or female, aged 18 through 75 years.
* If female, have a negative result from a serum pregnancy test at screening and a negative result from a serum or urine pregnancy test on Day -1.
* If male, agree to use an effective method of contraception (i.e., condom plus diaphragm with spermicide or condom plus spermicide) and not have their partners become pregnant throughout the study, or have been sterilized for at least 1 year (with supporting documentation of the absence of sperm in the ejaculate postvasectomy).
* If female of childbearing potential, agree to use an effective method of contraception (i.e., condom plus diaphragm with spermicide, condom plus spermicide, or nonhormonal intrauterine device) and not become pregnant throughout the study. Females who are at least 2-years postmenopausal (with supporting documentation from an obstetrician/gynecologist) or who have had tubal ligation or hysterectomy (with supporting documentation from the physician who performed the surgery) will not be considered to be of childbearing potential.
* Be nonsmoking (never smoked or have not smoked within the previous 2 years) or light smokers (less than or equal to 10 cigarettes per day within the previous 3 months).
* Have a sitting pulse rate greater than or equal to 50 beats per minute (bpm) or less than or equal to 100 bpm during the vital sign assessment at screening.
* Have a body mass index (BMI) greater than or equal to 18 kilograms per square meter and less than or equal to 42 kilograms per square meter.

Participants with Renal Impairment:

* Have results of medical history, physical examination, and laboratory and other test results consistent with their degree of renal impairment, as determined by the Investigator.
* Have an estimated glomerular filtration rate (eGFR) of 60-89 mL/min/1.73m2 (Group I); 30-59 mL/min/1.73m2 (Group II); and 15-29 mL/min/1.73 m2 (Group III). The maximum allowable intra-subject variability based on the 2 determinations of eGFR at screening and Day -1 using the Modification of Diet in Renal Disease (MDRD) equation is +/- 30%. If eGFR falls in different categories at screening and on Day -1, the Day -1 eGFR will be used for assignment to the renal impaired group.
* If receiving concomitant medications to treat underlying diseases or medical conditions related to renal insufficiency, must be on stable dosages of these medications for at least 8 weeks before screening.

Participants with Normal Renal Function:

- Have an eGFR greater than or equal to 90 mL/min/1.73 m2 at screening and on Day -1. The maximum allowable intra-subject variability based on the 2 determinations of eGFR at screening and Day -1 using the MDRD equation is +/- 30 percent. If eGFR falls in different categories at screening and Day -1, the Day -1 eGFR will be used to assign participant to study group.

Exclusion Criteria:

Common criteria:

* Known hypersensitivity to cebranopadol or other opioids.
* Abnormal ECG results thought to be potentially clinically significant according to the Investigator, or QT prolongation (QTcF greater than or equal to 450 msec; uncorrected QT greater than 500 msec).
* Positive test results for anti-human immunodeficiency virus type 1, hepatitis B surface antigen, hepatitis B core antibodies, or anti-hepatitis C virus at screening.
* History of alcohol or other substance abuse within the previous 5 years.
* Positive test results for benzoylecgonine (cocaine), methadone, barbiturates, amphetamines, benzodiazepines, alcohol, cannabinoids, opiates, or phencyclidine at screening or Day -1.
* Participation in any other clinical investigation using an experimental drug requiring repeated blood or plasma draws within 60 days of investigational product (IP) administration.
* Participation in a blood or plasma donation program within 60 or 30 days, respectively, of IP administration.
* Consumption of caffeine within 48 hours or consumption of alcohol within 72 hours before administration of IP.
* Consumption of beverages or food containing quinine (bitter lemon, tonic water) or any grapefruit-containing products, Seville oranges, or poppy seeds within 14 days before administration of IP.
* Any clinical condition or previous surgery that might affect the absorption, distribution, biotransformation, or excretion of cebranopadol.
* Employee, or immediate relative of an employee, of Forest Laboratories, Inc., any of its affiliates or partners, or the study center.
* Previously taken cebranopadol or previously participated in an investigational study of cebranopadol, unless otherwise authorized by the sponsor.
* Breastfeeding.

Participants with Renal Impairment:

* Clinically significant disease state, in the opinion of the examining physician, in any body system (other than renal function impairment or concomitant conditions for participants in groups I-III). Medical history, physical examination findings, and abnormal findings on electrocardiogram (ECG) and laboratory analyses should be reviewed, and the participant judged acceptable for participation in this study by the Investigator and Forest Medical Monitor.
* Sitting systolic blood pressure (BP) greater than or equal to 165 mm Hg or less than or equal to 95 mm Hg or sitting diastolic BP greater than or equal to 90 mm Hg or less than or equal to 50 mm Hg at screening.
* Abnormal and clinically significant results on physical examination, medical history, serum chemistry, hematology, or urinalysis with the exception of findings that are related to the renal disease process.
* Have undergone renal transplantation or had renal carcinoma within 1 year before screening.
* Have any evidence of skin lesions, diabetic foot, clinically significant edema states not judged to be related to renal failure, peripheral arterial disease, or epilepsy. (Edema [1+ to 3+ pitting] is allowed).
* History of or risks for acute pancreatitis or exacerbation of pancreatitis.
* Have taken any concomitant medications, with the exception of those medications prescribed as standard therapy for renal disease or other stable concomitant conditions, including over-the-counter medications, within 14 days before IP administration or hormonal drug products (except thyroid supplements) within 30 days before IP administration.

Participants with Normal Renal Function:

* Clinically significant disease state, in the opinion of the examining physician, in any body system.
* Sitting systolic BP greater than or equal to 140 mm Hg or less than or equal to 90 mm Hg or sitting diastolic BP greater than or equal to 90 mm Hg or less than or equal to 50 mm Hg at screening.
* Abnormal and clinically significant results on physical examination, medical history, oxygen saturation, serum chemistry, hematology, or urinalysis.
* Taken any concomitant medications (including over-the-counter medications) within 14 days or hormonal drug products (except thyroid supplements) within 30 days before administration of IP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2014-09-17 (Actual); Study Completion 2014-09-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter Plasma: maximum plasma concentration (Cmax) for Cebranopadol (GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Cmax was calculated based on plasma concentration-time data (using actual blood sampling times).
Pharmacokinetic parameter Plasma: maximum plasma concentration (Cmax) for M2 (7-hydroxy GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Cmax was calculated based on plasma concentration-time data (using actual blood sampling times).
Pharmacokinetic parameter Plasma: maximum plasma concentration (Cmax) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Cmax was calculated based on plasma concentration-time data (using actual blood sampling times).
Pharmacokinetic parameter Plasma: maximum plasma concentration (Cmax) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. Cmax was calculated based on plasma concentration-time data (using actual blood sampling times).
Pharmacokinetic parameter Plasma: time to maximum plasma concentration (tmax) for Cebranopadol (GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The time to maximum cebranopadol and its metabolites plasma concentration was calculated based on plasma concentration-time data (using actual blood sampling times).
Pharmacokinetic parameter Plasma: time to maximum plasma concentration (tmax) for M2 (7-hydroxy GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The time to maximum cebranopadol and its metabolites plasma concentration was calculated based on plasma concentration-time data (using actual blood sampling times).
Pharmacokinetic parameter Plasma: time to maximum plasma concentration (tmax) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The time to maximum cebranopadol and its metabolites plasma concentration was calculated based on plasma concentration-time data (using actual blood sampling times).
Pharmacokinetic parameter Plasma: time to maximum plasma concentration (tmax) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The time to maximum cebranopadol and its metabolites plasma concentration was calculated based on plasma concentration-time data (using actual blood sampling times).
Pharmacokinetic parameter Plasma: area under the plasma concentration-time curve from 0 to time t (AUC0-t) for Cebranopadol (GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-t was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: area under the plasma concentration-time curve from 0 to time t (AUC0-t) for M2 (7-hydroxy GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-t was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: area under the plasma concentration-time curve from 0 to time t (AUC0-t) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-t was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: area under the plasma concentration-time curve from 0 to time t (AUC0-t) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-t was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: the half-life associated with the terminal elimination phase (t1/2,z) for Cebranopadol (GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The half-life associated with the terminal elimination phase was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: the half-life associated with the terminal elimination phase (t1/2,z) for M2 (7-hydroxy GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The half-life associated with the terminal elimination phase was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: the half-life associated with the terminal elimination phase (t1/2,z) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The half-life associated with the terminal elimination phase was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: the half-life associated with the terminal elimination phase (t1/2,z) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The half-life associated with the terminal elimination phase was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: area under the plasma concentration-time curve extrapolated to infinity (AUC0-inf) for Cebranopadol (GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-inf was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: area under the plasma concentration-time curve extrapolated to infinity (AUC0-inf) for M2 (7-hydroxy GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-inf was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: area under the plasma concentration-time curve extrapolated to infinity (AUC0-inf) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-inf was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: area under the plasma concentration-time curve extrapolated to infinity (AUC0-inf) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC0-inf was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: extrapolated part of area under the plasma concentration-time curve (AUCt-inf) for Cebranopadol (GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUCt-inf was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: extrapolated part of area under the plasma concentration-time curve (AUCt-inf) for M2 (7-hydroxy GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUCt-inf was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: extrapolated part of area under the plasma concentration-time curve (AUCt-inf) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUCt-inf was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: extrapolated part of area under the plasma concentration-time curve (AUCt-inf) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUCt-inf was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: extrapolated AUC expressed as a percentage of total AUC0-inf (AUC%extr) for Cebranopadol (GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC%extr was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: extrapolated AUC expressed as a percentage of total AUC0-inf (AUC%extr) for M2 (7-hydroxy GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC%extr was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: extrapolated AUC expressed as a percentage of total AUC0-inf (AUC%extr) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC%extr was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: extrapolated AUC expressed as a percentage of total AUC0-inf (AUC%extr) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The AUC%extr was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: apparent clearance after oral administration (CL/f) for Cebranopadol (GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The CL/f was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Plasma: apparent volume of distribution after oral administration (Vz/f) for Cebranopadol (GRT6005) | Pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96, 120 and 168 hours post-dose
  PK blood samples were collected before administration of the IMP and for 168 hours after dosing; 18 PK blood samples were obtained from each participant. Plasma concentrations for cebranopadol were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Vz/f was calculated based on plasma concentration-time data (using the actual blood sampling times).
Pharmacokinetic parameter Urine: cumulative amount of unchanged drug excreted into the urine from time 0 to time t (Ae0-t) for Cebranopadol (GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae0-t was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: cumulative amount of unchanged drug excreted into the urine from time 0 to time t (Ae0-t) for M2 (7-hydroxy GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae0-t was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: cumulative amount of unchanged drug excreted into the urine from time 0 to time t (Ae0-t) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae0-t was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: cumulative amount of unchanged drug excreted into the urine from time 0 to time t (Ae0-t) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae0-t was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: cumulative amount of unchanged drug excreted into the urine from time 0 to time t expressed as a percentage of the dose (Ae%0-t) for Cebranopadol (GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae%0-t was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: cumulative amount of unchanged drug excreted into the urine from time 0 to time t expressed as a percentage of the dose (Ae%0-t) for M2 (7-hydroxy GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae%0-t was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: cumulative amount of unchanged drug excreted into the urine from time 0 to time t expressed as a percentage of the dose (Ae%0-t) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae%0-t was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: cumulative amount of unchanged drug excreted into the urine from time 0 to time t expressed as a percentage of the dose (Ae%0-t) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The Ae%0-t was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: renal clearance of drug from plasma (CLR) for Cebranopadol (GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The CLR was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: renal clearance of drug from plasma (CLR) for M2 (7-hydroxy GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The CLR was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: renal clearance of drug from plasma (CLR) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The CLR was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: renal clearance of drug from plasma (CLR) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The CLR was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: rate of renal excretion within collection period ti - tj (r) for Cebranopadol (GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The r was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: rate of renal excretion within collection period ti - tj (r) for M2 (7-hydroxy GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The r was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: rate of renal excretion within collection period ti - tj (r) for M3 (N-desmethyl-GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The r was calculated based on urine concentration-time data (using the actual urine sampling time intervals).
Pharmacokinetic parameter Urine: rate of renal excretion within collection period ti - tj (r) for M6 (7-hydroxy N-desmethyl-GRT6005) | Pre-dose and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 , and 96-120 hours intervals post-dose
  10 PK urine samples were obtained from each participant. Urine concentrations for cebranopadol and its metabolites were determined using validated high-performance liquid chromatography-tandem mass spectrometry bioanalytical assays. The r was calculated based on urine concentration-time data (using the actual urine sampling time intervals).

SECONDARY OUTCOMES:
Safety and tolerability of Cebranopadol (GRT6005): Number of participants with treatment emergent adverse events | Day 1 to Day 8
  Number of participants with treatment emergent adverse events. Treatment emergent adverse events were collected from dosing of IMP up to Day 8.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director Grünenthal GmbH, Study Director — Grünenthal GmbH
Locations (2):
- United States (2):
  - US0001 Contract research organization, Miami, Florida
  - US0002 Contract research organization, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No